CLINICAL TRIAL: NCT07054034
Title: A Randomized, Double-Blind, Placebo-Controlled Phase II Clinical Trial of MG-ZG122 Humanized Monoclonal Antibody Injection in Adult Subjects With Moderate-to-Severe Asthma to Evaluate Efficacy and Safety
Brief Title: Study of MG-ZG122 Humanized Monoclonal Antibody in Asthma Subjects
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Mabgeek Biotech.Co.Ltd (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MG-ZG122-AS-001
Record Dates: First submitted 2025-05-27; First posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Bronchial Asthma
Keywords: Bronchial Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Intervention Model Description: A Randomized, Double-Blind, Placebo-Controlled Phase II Clinical Trial of MG-ZG122 Humanized Monoclonal Antibody Injection in Adult Subjects with Moderate-to-Severe Asthma to Evaluate Efficacy and Safety
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- MG-ZG122 Regimen 1 (Experimental): Group MG-ZG122 210 mg Q12W: Subcutaneous injection of MG-ZG122 210 mg + subcutaneous injection of 2.0 mL placebo (to maintain blinding), administered once every 12 weeks, with a total of 4 administrations.
  Interventions: Drug: MG-ZG122 Humanized Monoclonal Antibody Injection
- MG-ZG122 Regimen 2 (Experimental): MG-ZG122 210 mg administered via subcutaneous injection plus 2.0 mL placebo via subcutaneous injection (to maintain blinding), once every 24 weeks. To maintain blinding, 4.0 mL placebo injections will be administered at Weeks 12 and 36, for a total of 4 doses.
  Interventions: Drug: MG-ZG122 Humanized Monoclonal Antibody Injection
- MG-ZG122 Regimen 3 (Experimental): MG-ZG122 420 mg administered via subcutaneous injection, once every 24 weeks. To maintain blinding, 4.0 mL placebo injections will be administered at Weeks 12 and 36, for a total of 4 doses.
  Interventions: Drug: MG-ZG122 Humanized Monoclonal Antibody Injection
- Placebo (Placebo Comparator): Subcutaneous injection of 0 mg (4.0 mL placebo) once every 12 weeks, for a total of 4 administrations.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: MG-ZG122 Humanized Monoclonal Antibody Injection — MG-ZG122 Humanized Monoclonal Antibody Injection
  Arms: MG-ZG122 Regimen 1; MG-ZG122 Regimen 2; MG-ZG122 Regimen 3
Other: Placebo — MG-ZG122 Humanized Monoclonal Antibody Injection Placebo
  Arms: Placebo

SUMMARY:
A Randomized, Double-Blind, Placebo-Controlled Phase II Clinical Trial to Evaluate the Efficacy and Safety of MG-ZG122 Humanized Monoclonal Antibody Injection in Asthma Subjects, with Dosing Every 12 or 24 Weeks for 48 Weeks

DETAILED DESCRIPTION:
This study is a multicenter, randomized, double-blind, placebo-controlled Phase II study. Approximately 160 adult asthma subjects are scheduled to receive multiple subcutaneous injections (every 12 or 24 weeks for 48 weeks). The study is divided into a screening period (1 week), a run-in period (4 weeks), a treatment period (48 weeks), and a follow-up period (12 weeks).

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following criteria to be enrolled in this study:

Age: 18 to 75 years old (inclusive), male or female.

Asthma Diagnosis:

Diagnosed with asthma for at least 1 year, and current disease status meets the diagnostic criteria of the 2024 GINA Guidelines (Global Initiative for Asthma).

Additionally:

Has received moderate-to-high dose inhaled corticosteroids (ICS) for at least 2 consecutive months prior to screening.

Pre-bronchodilator FEV1 (forced expiratory volume in 1 second) at screening and baseline visits is ≤80% of predicted normal value.

Asthma Control Questionnaire-5 (ACQ-5) score ≥1.5 at screening and baseline visits.

Has experienced ≥1 severe asthma exacerbation within the 12 months prior to screening.

Exclusion Criteria:

* 1， Known hypersensitivity to the investigational product or its excipients. 2，Clinical diagnosis of chronic obstructive pulmonary disease (COPD) or other lung diseases potentially impairing lung function (e.g., idiopathic pulmonary fibrosis, pneumothorax, atelectasis, pulmonary fibrosis, bronchial dysplasia, etc.), as determined by the investigator., 3，Experienced a severe asthma exacerbation during the screening period or within 1 month prior to dosing., 4，Received systemic glucocorticoid therapy from 1 month prior to screening to prior to dosing (excluding topical, ophthalmic, or intranasal glucocorticoids).

  5，Had pulmonary or other site infections requiring intravenous antibiotics, antifungal, or antiviral medications within 1 month prior to dosing.

  6，Received intravenous immunoglobulin (IVIG) therapy or allergen-specific immunotherapy (SIT) within 3 months prior to dosing.

  7，Used traditional Chinese herbal medicines with bronchodilatory or anti-asthmatic effects (excluding topical preparations) within 1 month prior to dosing.

  8，Underwent major surgery within 8 weeks prior to screening or planned to undergo major surgery during the study period (including hospitalized surgery and day-case surgery).

Ages: 15 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-05-11 (Actual); Primary Completion 2026-05-26 (Estimated); Study Completion 2027-05-26 (Estimated)

PRIMARY OUTCOMES:
Annual incidence rate of asthma exacerbations | 48week
  Annualized rate of severe asthma exacerbations over 48 weeks of treatment with MG-ZG122 compared to placebo.

SECONDARY OUTCOMES:
Absolute change in FEV1 from baseline | 12week
  Absolute change in pre-bronchodilator FEV1 from baseline at Week 12
Absolute change in FEV1 from baseline | 24week
  Absolute change in pre-bronchodilator FEV1 from baseline at Week 2424
Hospitalization due to asthma exacerbation events | 48week
  Annualized rate of hospitalizations or emergency department treatments due to severe asthma exacerbations during 48 weeks of treatment
Proportion of subjects with asthma exacerbations | 48week
  Proportion of subjects who experienced asthma exacerbations during 48 weeks of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- China-Japan Friendship Hospital, Beijing, China, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No